CLINICAL TRIAL: NCT06614894
Title: An Open Label Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacologic Properties of High Dose Ambroxol Hydrochloride in Adult (≥ 18 Years of Age) Subjects With MPS III
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ozlem Goker-Alpan (Other)
Collaborators: Team Sanfilippo (Unknown)
Responsible Party: Sponsor-Investigator, Ozlem Goker-Alpan, Principal Investigator, Lysosomal and Rare Disorders Research and Treatment Center, Inc.
Organization: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-LDRTC-01
Record Dates: First submitted 2024-08-28; First posted 2024-09-26 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-09

CONDITIONS: Sanfilippo Syndrome; MPS3
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Tablets; Ambroxol

STUDY DESIGN:
Intervention Model Description: A Non-randomized (single arm) clinical trial where all participants will receive the same experimental therapy and undergo the same dose escalation plan. All participants will be followed over time to observe their response related to safety and effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ambroxol Hydrochloride 30mg - 9mg/kg/day (Experimental): Ambroxol Hydrochloride 30mg Dose escalation: Initial dose of 9mg/kg/day (or max dose 150mg TID)
  Interventions: Drug: Ambroxol Hydrochloride 30 mg tablet - 9 mg/kg/day
- Ambroxol Hydrochloride 30mg - 18mg/kg/day (Experimental): Ambroxol Hydrochloride 30mg Dose escalation: 18mg/kg/day (or max dose 300mg TID)
  Interventions: Drug: Ambroxol Hydrochloride 30 mg tablet - 18 mg/kg/day
- Ambroxol Hydrochloride 30mg - 27mg/kg/day (Experimental): Ambroxol Hydrochloride 30mg Dose escalation: 27mg/kg/day (or max dose 1350mg QD)
  Interventions: Drug: Ambroxol Hydrochloride 30 mg tablet - 27 mg/kg/day

INTERVENTIONS:
Drug: Ambroxol Hydrochloride 30 mg tablet - 9 mg/kg/day — Ambroxol Hydrochloride 30 mg oral pill/tablet - 9 mg/kg/day
  Other Names: Ambroxol
  Arms: Ambroxol Hydrochloride 30mg - 9mg/kg/day
Drug: Ambroxol Hydrochloride 30 mg tablet - 18 mg/kg/day — Ambroxol Hydrochloride 30 mg oral pill/tablet - 18 mg/kg/day
  Other Names: Ambroxol
  Arms: Ambroxol Hydrochloride 30mg - 18mg/kg/day
Drug: Ambroxol Hydrochloride 30 mg tablet - 27 mg/kg/day — Ambroxol Hydrochloride 30 mg oral pill/tablet - 27 mg/kg/day
  Other Names: Ambroxol
  Arms: Ambroxol Hydrochloride 30mg - 27mg/kg/day

SUMMARY:
A dose escalation study to evaluate the safety, tolerability, and pharmacologic properties of Ambroxol in adult participants with Sanfilippo disease(s) (MPS3).

DETAILED DESCRIPTION:
This is a dose escalation study in which open label Ambroxol 30mg (study drug) will be administered to adult patients with Sanfilippo Disease (MPS3). Administration route of study drug will be either crushed and mixed with soft foods or as an Ambroxol suspension through a feeding tube, if applicable.

Study Timeline - Screening: 4 weeks (28 days) Treatment Period: 52 weeks Post-Treatment (after Week 52): 4 weeks withdrawal/safety follow-up period

Patients will be screened at which point a thorough review of the Informed Consent form will be completed, sNFL levels, urinary GAGs, and serum HS results/data from the previous 12 months will be reviewed, urine and blood will be collected, complete questionnaires, Motor skills assessments, and evaluation by the Principal Investigator (PI).

Eligible patients will proceed to receive the initial Ambroxol dose of 9mg/kg/day (maximum dose of 150 mg TID) divided into three equal doses per day, on-site. Other assessments including blood and urine collection, ECG, motor skills assessments, hearing test, questionnaires, and evaluation by the PI will be completed.

Following the first day of dosing, a virtual visit will be performed via Telemedicine within 1 week of dose start to assess safety.

At Weeks 12 and 24, enrolled patients will return to site for Ambroxol dose escalation to 18mg/kg/day (max dose of 300 mg TID) and 27mg/kg/day (max dose of 1350 mg/day), respectively. Assessments including blood and urine collection, ECG, motor skills assessments, hearing test, questionnaires, and evaluation by the PI will be completed at these visits.

Telemedicine visits will take place at Weeks 13 and 25, to assess safety.

At Week 36, a safety visit will be performed in which blood and urine will be collected.

At Week 52, end of study assessments will be completed which includes blood and urine collection, motor skills assessments, hearing test questionnaires, and evaluation by the PI will be conducted and treatment will be stopped.

A safety follow-up visit will be done 4 weeks after Week 52 visit is completed in which the patient will be evaluated by the PI.

ELIGIBILITY:
Inclusion Criteria:

1. IRB - approved informed consent/assent signed by subject and/or parent(s) or legal guardian(s).
2. Genetically confirmed diagnosis of MPS III disease.
3. Genomic DNA analysis demonstrating a homozygous or compound heterozygous pathogenic variants in SGSH (type A), NAGLU (type B), HGSNAT (type C), or GNS (type D) genes. Type E will not be studied.
4. Elevated excretion of urinary GAGs and/or serum HS (if no historical data is available, screening GAGs and serum HS values will be utilized to assess inclusion criteria).
5. Male or female; eighteen years of age and older, who is able to take Ambroxol Hydrochloride orally.
6. Negative urine pregnancy test at screening for female subjects with child-bearing potential.
7. The subject is willing to abstain from consumption of grapefruit, grapefruit juice, or grapefruit containing products for 72 hours prior to administration of the first dose of Ambroxol and for the duration of the treatment period.

Exclusion Criteria:

1. Unwilling or unable to follow protocol requirements as per principal investigator.
2. Any serious or chronic medical illness, including significant cardiac or severe debilitating pulmonary disease.
3. Poorly controlled seizures, defined as more than one seizure per day for the past 6 months.
4. Medications identified as a strong inducers or inhibitors of CYP3A, and changing to another alternative drug to treat the condition would place the subject at undue risk.
5. Any medical condition that, in the opinion of the PI, would make the subject unsuitable to participate in the study.
6. Inability to cooperate for clinical and safety data collection.
7. Known hypersensitivity to Ambroxol or any of its excipients.
8. Use of genistein or Miglustat within one week of starting screening.
9. Evidence of hepatitis B or hepatitis C infection upon serological testing at screening.
10. Currently participating in another clinical trial or has completed an interventional trial less than 2 weeks prior to screening visit.
11. The subject has received strong inducers (Note: eg, herbal supplements) or inhibitors of CYP3A within 15 days or 5 half-lives from screening, whichever is longer, prior to enrollment. This also includes the consumption of grapefruit, grapefruit juice, or grapefruit containing products within 72 hours of starting Ambroxol administration.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | From baseline to 52 weeks
  1. Safety and tolerability as measured by number of Participants with at least one serious and at least one non-serious Treatment Emergent Adverse Events (TEAEs), assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Changes in physical examination from baseline in motor capabilities and disease state: Physician (Clinician) Global Impression of Change | From baseline to 52 weeks
  Physician (Clinician) Global Impression of Change (scale: 0-very much worse - 7-Very much improved).
Change from baseline in EQ-5D-5L™ or EQ-5D-Y™ | From baseline to 52 weeks
  Change from baseline in EQ-5D-5L™ or EQ-5D-Y™
Change from baseline in VABS-III age equivalent scores (AEqs) | From baseline to 52 weeks
  Vineland Adaptive Behavior scale-III
Assessment of Pharmacokinetics of Ambroxol in subjects with MPS III | From baseline to 52 weeks
  Plasma PK parameter estimates for oral Ambroxol include the area under the curve (AUC).
Assessment of Pharmacokinetics of Ambroxol in subjects with MPS III | From baseline to 52 weeks
  Plasma PK parameter estimates for oral Ambroxol include maximum concentration (Cmax).
Assessment of Pharmacokinetics of Ambroxol in subjects with MPS III | From baseline to 52 weeks
  Plasma PK parameter estimates for oral Ambroxol include time to maximum dose concentration (Tmax).
Assessment of Pharmacokinetics of Ambroxol in subjects with MPS III | From baseline to 52 weeks
  Plasma PK parameter estimates for oral Ambroxol include terminal half-life (t1/2).
Assessment of Pharmacodynamics of Ambroxol in subjects with MPS III | From baseline to 52 weeks
  Changes from baseline in Urinary GAG levels as measured by total quantified concentration. Changes from baseline will be analyzed using main effects, fixed for treatment (dose), categorical visit number, treatment-by-visit interaction, baseline value as covariate, and subject as the random effect.
Assessment of Pharmacodynamics of Ambroxol in subjects with MPS III | From baseline to 52 weeks
  Serum Heparan sulfate (HS) level changes from baseline as measured by total quantified concentration. Changes from baseline will be analyzed using main effects, fixed for treatment (dose), categorical visit number, treatment-by-visit interaction, baseline value as covariate, and subject as the random effect.
Change from baseline in Timed up and go (TUG) test | From baseline to 52 weeks
  Change from baseline in Timed up and go (TUG) test and in ABR at Week 52 may also be tested for correlations.
Change from baseline in 10-meter walk test | From baseline to 52 weeks
  Change from baseline in 10-meter walk test, may also be tested for correlations.
Change from baseline in SBRS | From baseline to 52 weeks
  Change from baseline in SBRS

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — Lysosomal & Rare Disorders Research & Treatment Center, Inc.
Locations (1):
- Lysosomal & Rare Disorders Research & Treatment Center, Inc., Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No